CLINICAL TRIAL: NCT03241485
Title: Randomized, Double Blinded, Trial Comparing Intrathecal Morphine With Placebo in Patients Undergoing Robotic Totally Endoscopic Beating Heart Coronary Revascularization and Intraoperative Extubation
Brief Title: Trial Comparing Intrathecal Morphine With Placebo In Patients Undergoing Robotic Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB17-1103
Record Dates: First submitted 2017-05-20; First posted 2017-08-07 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into 2 groups. The placebo group will receive intrathecal saline. The morphine group will receive intrathecal morphine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will receive intrathecal intervention and will not know which group they are assigned to. The provider performing the procedure and collecting the data will also be blinded to the intervention assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 60 patients will be randomly assigned to this arm. The patients in this arm will receive intrathecal saline.
  Interventions: Drug: Placebo
- Intrathecal morphine (Active Comparator): 60 patients will be randomly assigned to this arm. The patients in this arm will receive intrathecal morphine.
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Intrathecal morphine — 5 micrograms/kilogram of intrathecal morphine administered in the spinal space, not to exceed 1mg
  Other Names: Duramorph
  Arms: Intrathecal morphine
Drug: Placebo — Saline intrathecal given in the same manner as the intervention groups.
  Arms: Placebo

SUMMARY:
This is a randomized clinical trial in patients undergoing robotic myocardial revascularization with intraoperative extubation. Patients will be randomized into placebo or intrathecal morphine groups to assess postoperative pain scores and patient satisfaction. Patients will also be assessed for side effects from the intervention.

DETAILED DESCRIPTION:
Following Institutional Review Board approval and informed patient consent, 120 patients scheduled for elective robotic myocardial revascularization without cardiopulmonary bypass and anticipated intraoperative tracheal extubation will be studied. Patients will be randomized into one of two groups. Group A (placebo, control group) will receive intrathecal normal saline, Group B (morphine group) intrathecal morphine. All procedures will occur and administered medications given immediately prior to induction of general anesthesia in the operating room. Power analysis indicates that 60 patients per Group is appropriate, as further described below. Inclusion criteria include any patient undergoing elective robotic myocardial revascularization without anticipated use of cardiopulmonary bypass and with anticipated intraoperative tracheal extubation. Exclusion criteria include emergency surgery, ejection fraction less than 40%, preoperative use of inotropic agents or intraaortic balloon pump, anticipated use of cardiopulmonary bypass, previous cardiothoracic surgery, anticipated postoperative tracheal intubation, severe pulmonary disease, morbid obesity (BMI >35 kg/m2), severe renal dysfunction (creatinine > 1.5) recent history of opioid abuse, preoperative use of opioids, or any contraindication to intrathecal injection (patient refusal, difficult patient anatomy, pre-existing coagulopathy, morphine allergy).

Routine preoperative data will be collected (see Preoperative Data Sheet). Following intravenous access and routine mild sedation, each patient will be transported to the operating room and assume the sitting position. Following routine skin preparation, a routine lumbar intrathecal injection will be made via a 22-g spinal needle. The injectate will be either morphine (5 mcg/kg, maximum dose of 1 mg) or normal saline. The injectate will be prepared by a co-Investigator not directly involved in patient care. Thus, all preoperative, intraoperative, and postoperative caregivers will be blinded to intrathecal injectate composition (all injectates will be standardized to a total of 1.0 ml). All patients will have port incisions injected with 60 ml of 0.25% bupivacaine by the surgeon after the completion of surgery.

Following intrathecal injection, the patient will then assume the supine position. An arterial catheter will be inserted and general endotracheal anesthesia will be induced. Intraoperative anesthetic technique will be standardized and equivalent between Groups (see Intraoperative Anesthetic Protocol Sheet). The anesthetic protocol will allow tracheal extubation to occur in the operating room immediately after surgery (if clinically indicated).

Surgical technique will not be altered in any way. All patients in both Groups will be operated on by the same surgeon. Routine intraoperative data will be collected (see Intraoperative Data Sheet). In all patients, tracheal extubation will be attempted in the operating room immediately after surgery (if clinically indicated).

Both Groups will receive routine postoperative care and identical postoperative analgesic protocols to assess adequacy of postoperative analgesia (see Postoperative Analgesia Protocol and Postoperative Data Sheets). The American Pain Society Outcome Questionnaire (APS-POQ) will be administered to patients prior to discharge (see data sheet).15

ELIGIBILITY:
Inclusion Criteria:

• patient undergoing elective robotic myocardial revascularization without anticipated use of cardiopulmonary bypass and with anticipated intraoperative tracheal extubation.

Exclusion Criteria:

* Emergency surgery
* Preoperative use of inotropes/IABP
* Preoperative use of opoids
* Ejection fraction less than 40%
* Anticipated use of cardiopulmonary bypass
* Previous cardiothoracic surgery
* Anticipated postoperative tracheal intubation
* severe pulmonary disease
* morbid obesity (BMI >35 kg/m2)
* severe hepatic impairment
* severe renal dysfunction (creatinine > 1.5)
* any contraindication to intrathecal injection (patient refusal, difficult patient anatomy, pre-existing coagulopathy, morphine allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richa Dhawan, MD, MPH, Principal Investigator — University of Chicago Hospital
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 42 patients were randomized to the intrathecal placebo group. This group received a normal saline injected in the spinal spice, prior to surgery.
- Intrathecal Morphine: 37 patients were randomized to the intrathecal morphine group. This group received 5 micrograms/kilogram of intrathecal morphine administered in the spinal space
Period: Overall Study
Arm/Group | Placebo | Intrathecal Morphine
Started | 42 | 37
Completed | 37 | 33
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 42 patients were randomized to this group
- Intrathecal Morphine: 37 patients were randomized to this group
- Total: Total of all reporting groups
Arm/Group | Placebo | Intrathecal Morphine | Total
Number analyzed (Participants) | 42 | 37 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10) | 67.3 (10.5) | 65.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 33 | 32 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: KG] | 87 (14) | 85 (14) | 86.4 (14.2)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.6 (3.6) | 27.5 (3.2) | 28 (3.3)
ASA Physical Status [Median (Inter-Quartile Range); unit: Units on a scale] — ASA Physical status is a medical grading system in which it can help predict a patients perioperative risks. The higher the number, the most at risk the patient is and possibility of a worse outcome. ASA grading scale Ranges from 1-6
  Units on a scale | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]
EuroSCORE II [Mean (Standard Deviation); unit: Scores on a scale] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) II. Predicts risk of in-hospital mortality after major cardiac surgery. This is calculated on a score on a scale by entering several different information of the patient into the Euroscore II calculator. These include demographic, lab values, medical history.
  The higher a patients total score is, the likelihood of post-operative mortality after cardiac surgery is. With a range from 0-21. With 0 meaning there there is no risk of in-hospital mortality after major cardiac surgery and 21 meaning there is a severe high risk.
  Scores on a scale | 1 (0.5) | 1 (0.5) | 1 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Morphine Consumption
Description: We anticipate that patients in the intervention groups will require less postoperative morphine for pain control.
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Miligram
Groups:
- Placebo: 36 patients were analyzed for primary outcome. One patient did not receive allocated intervention (failed spinal), One PCA data was lost, and 4 patients remained intubated overnight.
- Morphine: Intrathecal morphine group
Arm/Group | Placebo | Morphine
Number analyzed (Participants) | 36 | 33
Miligram | 59 [41 to 79] | 28 [16 to 46]

2. Secondary Outcome: Pain Score
Description: Patients will score their pain on a visual analog scale of 0-10. The higher the score, the worse the patients reported pain is at that time .
Time Frame: First 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Placebo: Intrathecal saline group
Arm/Group | Placebo | Morphine
Number analyzed (Participants) | 37 | 33
score on a scale | 6 [4.5 to 8] | 1.2 [0 to 2.5]

3. Secondary Outcome: Patient Satisfaction
Description: Patients will take a satisfaction survey prior to discharge, this is measured by calculating a score on a scale. This survey consist of questions that asks about the subjects post-operative experience with pain. Higher reported scores represent worse post-operative subject experience. These are ranked from a 0-10 scale, where 0 is the best experience and 10 meaning the worst experience. Questions being asked how satisfied they were with the results of the pain treatment while hospitalized, least pain in prior 24 hours, worst pain in prior 24 ours, percent time in severe pain, how much pain interfered with different activities, how much pain caused anxiety, depression, fright, helplessness, how severe were symptoms of nausea, drowsiness, itching, dizziness, and percentage pain relief in prior 24 hours.
Time Frame: 1-3 days after surgery, prior to discharge.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Morphine
Number analyzed (Participants) | 28 | 35
score on a scale | 9 [7 to 10] | 9.5 [6.5 to 10]

4. Secondary Outcome: Number of Participants With Nausea
Description: Daily evaluation of nausea post-operatively throughout the subjects hospital stay.
Time Frame: Until discharge, 2-3 days after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Nausea): Intrathecal saline group
Arm/Group | Placebo (Nausea) | Morphine
Number analyzed (Participants) | 37 | 33
Participants | 3 | 12

5. Secondary Outcome: Number of Participants With Respiratory Depression
Description: Opioid related respiratory depression, post-operatively throughout the subjects hospital stay.
Time Frame: During hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Morphine
Number analyzed (Participants) | 37 | 33
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Each subject was assessed for adverse events throughout their hospital stay, on average this was 1-2 days per participant.
Groups:
- Morphine: 5 micrograms/kilogram of intrathecal morphine.
Arm/Group | Placebo | Morphine
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/37
Other Adverse Events (participants affected / at risk) | 0/42 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT03241485/Prot_SAP_001.pdf